CLINICAL TRIAL: NCT01156012
Title: Efficacy and Safety Assessment of T2345 in Ocular Hypertensive or Glaucomatous Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT2345-PIII-12/08; 2009-011157-41 (EudraCT Number)
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2014-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Prostaglandins

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- T2345 (Experimental): One drop of T2345
  Interventions: Drug: T2345
- Prostaglandin (Active Comparator): One drop
  Interventions: Drug: Prostaglandin

INTERVENTIONS:
Drug: T2345 — One drop of T2345
  Arms: T2345
Drug: Prostaglandin — One drop
  Arms: Prostaglandin

SUMMARY:
The purpose of this study is to assess the efficacy and safety of T2345 versus active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with glaucoma

Exclusion Criteria:

* Under 18.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Director, Clermont-Ferrand, France

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Included patients= 404 patients but 2 patients without available data after Day 0. These 2 patients were excluded from the analyses sets.
Groups:
- T2345: One drop of T2345
  T2345: One drop of T2345 at 9.00pm
- Prostaglandin: One drop of prostaglandin
  Prostaglandin: One drop of prostaglandin at 9.00pm
Period: Overall Study
Arm/Group | T2345 | Prostaglandin
Started | 213 | 189
Completed | 206 | 186
Not Completed | 7 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — use of commercial drug instead of study | 0 | 1
Not completed — Non respect of one of inclusion criteria | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety set
Groups:
- Total: Total of all reporting groups
Arm/Group | T2345 | Prostaglandin | Total
Number analyzed (Participants) | 213 | 189 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.4) | 65.7 (11.7) | 64.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 86 | 200
  Male | 99 | 103 | 202
Region of Enrollment [Number; unit: participants]
  France | 104 | 93 | 197
  Belgium | 14 | 8 | 22
  Italy | 25 | 22 | 47
  Spain | 8 | 7 | 15
  Portugal | 15 | 15 | 30
  Tunisia | 47 | 44 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: The worse eye is defined as:
  * If both eyes are eligible the eye with highest Intraocular pressure (IOP) at Day 0 (D0). If both eyes have the same IOP at D0 the worse eye is the right eye.
  * If only one eye is eligible this eye is the worse eye.
  * If neither eye is eligible the worse eye is defined as the eye with the highest IOP at D0.
  If both eyes have the same IOP at D0 the worse eye is the right eye.
Time Frame: Day 0 and Day 84
Population: mITT set : All randomised patients, with at least one eligible eye, having received at least one dose of the Investigational Medicinal Product, and for whom any follow-up IOP recording was available for the worse eye.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | T2345 | Prostaglandin
Number analyzed (Participants) | 189 | 164
mmHg | -8.6 (2.6) | -9.0 (2.4)

ADVERSE EVENTS:
Arm/Group | T2345 | Prostaglandin
Serious Adverse Events (participants affected / at risk) | 5/213 | 1/189
Other Adverse Events (participants affected / at risk) | 0/213 | 0/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T2345 (N=213) | Prostaglandin (N=189)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results of the Trial are the sole and exclusive property of THEA, and cannot be used in whatever form without prior written agreement of THEA.